CLINICAL TRIAL: NCT06661720
Title: Short TeRm Intensified Pembrolizumab (KEytruda) and Tivozanib for High-Risk Renal Cell Carcinoma - STRIKE
Brief Title: Testing the Addition of the Anti-Cancer Drug Tivozanib to Immunotherapy (Pembrolizumab) After Surgery to Remove All Known Sites of Kidney Cancer
Acronym: STRIKE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A032201; NCI-2024-08233 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Clear Cell Renal Cell Carcinoma; Renal Cell Carcinoma (RCC); Stage II Renal Pelvis Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; tivozanib; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV on days 1 and 43 of each cycle, or on days 1, 22, 43 and 64 of each cycle. Cycles repeat every 12 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI or CT throughout the trial and may undergo tissue biopsy on study.
  Interventions: Biological: Pembrolizumab; Procedure: Biospecimen Collection; Procedure: MRI; Procedure: Computed Tomography; Procedure: Biopsy; Other: Questionnaire Administration
- Arm 2 (pembrolizumab + tivozanib) (Experimental): Patients receive pembrolizumab IV on days 1 and 43 of each cycle and tivozanib PO QD on days 1-21, days 29-49, and days 57-77 of each cycle for up to 6 months. Cycles repeat every 12 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI or CT throughout the trial and may undergo tissue biopsy on study.
  Interventions: Biological: Pembrolizumab; Drug: Tivozanib; Procedure: Biospecimen Collection; Procedure: MRI; Procedure: Computed Tomography; Procedure: Biopsy; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Pembrolizumab — Given intravenously
  Other Names: Keytruda
Drug: Tivozanib — Given orally
  Arms: Arm 2 (pembrolizumab + tivozanib)
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: MRI — Undergo MRI
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CT Scan; CAT Scan
Procedure: Biopsy — Undergo biopsy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding tivozanib to standard therapy pembrolizumab versus pembrolizumab alone for the treatment of patients with high-risk renal cell carcinoma (RCC). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Tivozanib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals tumor cells to multiply. This helps stop the spread of tumor cells. Giving pembrolizumab and tivozanib together may work better than pembrolizumab alone in treating patients with RCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare disease free survival (DFS) as assessed by the investigator for high-risk renal cell carcinoma patients treated with adjuvant pembrolizumab and tivozanib versus those receiving pembrolizumab alone.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) for patients treated with adjuvant pembrolizumab and tivozanib versus those receiving pembrolizumab alone.

II. To assess adverse events in each study arm by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

BIOBANKING OBJECTIVE:

I. To bank specimens for future unspecified research.

QUALITY OF LIFE (QOL) OBJECTIVES:

I. To compare global quality of life (QOL) for patients treated with pembrolizumab and tivozanib versus those receiving pembrolizumab alone.

II. To compare patient-reported fatigue for patients treated with pembrolizumab and tivozanib versus those receiving pembrolizumab alone.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pembrolizumab intravenously (IV) on days 1 and 43 of each cycle, or on days 1, 22, 43 and 64 of each cycle. Cycles repeat every 12 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and magnetic resonance imaging (MRI) or computed tomography (CT) throughout the trial and may undergo tissue biopsy on study.

ARM II: Patients receive pembrolizumab IV on days 1 and 43 of each cycle and tivozanib orally (PO) once daily (QD) on days 1-21, days 29-49, and days 57-77 of each cycle for up to 6 months. Cycles repeat every 12 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and MRI or CT throughout the trial and may undergo tissue biopsy on study.

After completion of study treatment, patients are followed up every 4 months for 2 years, then every 6 months for 3 years, then every subsequent year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed diagnosis of RCC with clear cell component with or without sarcomatoid features following complete resection of the primary tumor (radical or partial nephrectomy)

  * Note: Patients with microscopically positive soft tissue or vascular margins without gross residual disease are permitted

    * Intermediate-high risk RCC:

      * pT2 grade 4 or sarcomatoid features, N0M0
      * pT3 any grade N0, M0
    * High-risk RCC

      * pT4, any grade, N0, M0
      * pT, any stage., any grade, N+, M0
    * cM1 no evidence of disease (NED) RCC

      * Participants who have had resection of primary tumor (radical or partical nephrectomy) and resection or definitive radiation or ablation of solid, isolated, soft tissue metastases (excluding brain and bone lesions) at the time of primary tumor removal (synchronous) or ≤1 year from primary tumor removal (metachronous)

        * Surgery (radical or partial nephrectomy or metastasectomy or ablation) > 4 weeks but =< 16 weeks prior to study registration with no ongoing complications from surgery
        * No evidence of disease at time of randomization as assessed by investigator by either CT or MRI scan of the brain and chest, abdomen and pelvis
        * No prior systemic treatment for RCC
        * Age >= 18 years
        * Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (or Karnofsky >= 60%)
        * Absolute neutrophil count (ANC) >= 1,000/mm^3
        * Platelet count >= 100,000/mm^3
        * Hemoglobin >= 8 g/dL
        * Total bilirubin =< 3 x upper limit of normal (ULN)
        * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN)
        * Calculated (calc.) creatinine clearance >= 30 mL/min (using Cockcroft Gault equation or the estimated glomerular filtration rate from the modification of diet in renal disease trial)
        * Urine protein =< 1+ on urine analysis (UA) or urine protein creatinine ration (UPCR) < 2mg/mg
        * Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative pregnancy test is required =< 14 days prior to registration
        * HIV status: HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
        * Hepatitis
  * Hepatitis B: For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with resolved HBV infection, defined as positive hepatitis B core antibody (anti-HBc) and negative hepatitis B surface antigen (HbsAg), are eligible
  * Hepatitis C: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load

    * Cardiac Disease: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class IIB or better
    * No history of myocarditis
    * No history of clinically significant pneumonitis
    * No uncontrolled hypertension (systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg) documented on 2 consecutive measurements taken at least 2 hours apart
    * No serious non-healing wound, ulcer or bone fracture within 28 days prior to registration
    * No serious/active infection requiring parenteral antibiotics
    * No moderate or severe hepatic impairment (child-Pugh B or C)
    * No significant bleeding disorders within 1 month prior to registration, for example:
  * Hematemesis, hematochezia or other gastrointestinal bleeding grade 3 or higher
  * Hemoptysis of pulmonary bleeding grade 3 or higher
  * Hematuria or other genitourinary bleeding grade 3 or higher

    * No history of allogeneic organ transplantation
    * No history of allergy of hypersensitivity to study drugs or components
    * No condition requiring systemic treatment with either corticosteroid (> 10 mg daily or prednisone equivalent) within 14 days of treatment initiation or other immunosuppressive medications within 30 days of randomization. Inhaled or topical steroids and adrenal replacement doses ≤10 mg daily prednisone equivalent are permitted in absence of active autoimmune disease
    * No active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis or other gastrointestinal condition associated with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 4 weeks prior to registration
    * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
    * No patients with a history of autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids > 10 mg/day, or immunosuppressive drugs) with the following exceptions:
  * Replacement therapy (e.g., thyroxine, insulin, physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
  * Brief (<7 days) use of systemic corticosteroids is allowed when use is considered standard of care
  * Patients with vitiligo, psoriasis, type 1 diabetes mellitus, hypothyroidism, or resolved childhood asthma/atopy will not be excluded
  * Patients requiring intermittent use of bronchodilators, inhaled steroids, or local steroid injections will not be excluded
  * Patients with hypothyroidism that is stable with hormone replacement or Sjögren's syndrome will not be excluded • Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2037-11 (Estimated); Study Completion 2037-11 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From time of randomization until disease recurrence or death, assessed up to 10 years
  The primary analysis will be a comparison of DFS between the two study arms using a stratified log-rank test. The treatment effect will be estimated with a hazard ratio (HR) and corresponding 95% confidence interval obtained from a stratified Cox model with treatment group (experimental group versus control group) as the explanatory variable. Interim analyses: There will be several futility analyses for the trial. These analyses will employ the linear 20% method proposed by Freidlin, Korn and Gray. Based on the current design parameters, the first analysis would be performed at 37% information (99 DFS events), and the trial would be stopped for futility if the observed hazard ratio (experimental versus [vs.] control) were worse than 1. Additional analyses will be performed at 50% (133 DFS events), 60% (159 DFS events), and 70% information (186 DFS events), the trial would be stopped for futility if the observed HR were worse than 0.983, 0.971 and 0.959, respectively.

SECONDARY OUTCOMES:
Overall survival (OS) | From time of randomization until death, assessed up to 10 years
  The OS will be compared between the two treatment arms using a stratified log-rank test. An estimate of the OS difference between the arms will be made with a HR generated by a stratified Cox model. A point estimate and 95% confidence interval will be generated. If there are clinically meaningful imbalances between the treatment arms, a secondary analysis for DFS will be performed with a multivariable Cox model that includes the stratification variable and all baseline variables with meaningful differences. A similar analysis will be done for the OS endpoint. Key subgroup analyses will be performed to determine whether there is evidence that the treatment effect differs among subgroups that correspond to key prognostic variables. This includes the stratification variable.
Incidence of adverse events (AEs) | From baseline to 10 years after registration
  These will be assessed using Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be summarized with frequencies and relative frequencies. The maximum grade for an AE will be recorded for each patient by treatment arm. The number (percent) of patients that experience each observed adverse event will be summarized by treatment arm. In addition, the proportion of patients that experience a grade 3+, grade 4+, and grade 5 adverse event will be summarized as the number and percent of patients by treatment arm. The primary summary will be regardless of attribution. Will also have an analogous summary for the adverse events that were deemed at least possibly related to treatment.
Proportion of patients that tolerate pembrolizumab and tivozanib | From day 1 to 6 months
  Tolerability will be defined as the ability of a patient to receive at least half the planned doses of tivozanib in combination with pembrolizumab if they have not had a DFS event. This will be determined as the number of patients on arm 2 who received at least one dose of tivozanib, who have not had a DFS within 6 months, and who received at half of the planned doses tivozanib divided by the number of patients on arm 2 who received at least one dose of tivozanib and who have not had a DFS within 6 months. The proportion of patients who tolerated tivozanib in combination with pembrolizumab will be estimated with a binomial point estimate and 95% binomial confidence interval.

OTHER OUTCOMES:
Estimates of treatment effect by sex | Up to 10 years
  Estimates of DFS and the corresponding 95% CIs will be evaluated by sex.
Estimates of treatment effect by race | Up to 10 years
  Estimates of DFS and the corresponding 95% CIs will be evaluated by race
Estimates of treatment effect by ethnicity | Up to 10 years
  Estimates of DFS and the corresponding 95% CIs will be evaluated by ethnicity.

CONTACTS AND LOCATIONS:
Locations (393):
- United States (393):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope Upland, Upland, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Hartford Healthcare - Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Outpatient Center - Oak Lawn, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - UPMC Western Maryland, Cumberland, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided